CLINICAL TRIAL: NCT01050101
Title: The Effect of Meal Viscosity on Postprandial Metabolic, Gut Hormone and Satiety Responses to Low and High Glycemic Index Preload Meals in Overweight Pre- and Post-menopausal Women.
Brief Title: The Effects of Fiber on Appetite and Digestion Hormones
Acronym: FS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FS 2009-052
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Psychological Phenomena and Processes; Nutrition Physiological Phenomena
Keywords: Satiety; Fiber; Nutrition; Pre- and post-menopausal women; overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- High GI low fiber meal (Placebo Comparator): No fiber control meal
  Interventions: Dietary Supplement: No fiber
- Low GI high fiber viscous meal (Active Comparator): 80:20 ratio of viscous polysaccharide fiber to insoluble non-viscous producing fiber
  Interventions: Dietary Supplement: Low GI high fiber viscous meal
- Low GI high fiber non-viscous meal (Active Comparator): 20:80 ratio of viscous polysaccharide fiber source to insoluble non-viscous producing fiber
  Interventions: Dietary Supplement: Low GI high fiber non-viscous

INTERVENTIONS:
Dietary Supplement: No fiber — The High GI low fiber meal consists of 0 grams fiber with total kcal of 573 with 63% energy from carbohydrates, 24% energy from fat and 13% energy from protein.
  Test meal consists of breakfast meals containing muffins and yogurt beverage/shake.
  Arms: High GI low fiber meal
Dietary Supplement: Low GI high fiber viscous meal — Test meal consists of 12 grams of fiber (9 grams soluble and 3 grams insoluble). The ratio is 80:20 ratio of viscous polysaccharide fiber source (psyllium husk) to insoluble non-viscous producing fiber source (cellulose).
  Total kcal provided as 560 kcal with 63% energy from carbohydrates, 24% energy from fat and 13% energy from protein. Test meal consists of breakfast meals containing muffins and yogurt beverage/shake.
  Arms: Low GI high fiber viscous meal
Dietary Supplement: Low GI high fiber non-viscous — Test meal consists of 11 grams of fiber (3 grams soluble and 8 grams insoluble). The ratio is 20:80 of viscous polysaccharide fiber source (psyllium husk) to insoluble non-viscous producing fiber source (cellulose).
  Total kcal provided as 560 kcal with 63% energy from carbohydrates, 24% energy from fat and 13% energy from protein. Test meal consists of breakfast meals containing muffins and yogurt beverage/shake.
  Arms: Low GI high fiber non-viscous meal

SUMMARY:
In this research study, investigators are interested in how certain dietary fibers in the diet affect certain hormones released from your intestine after eating and how these influence your appetite. The study hypothesis is that certain fibers will slow digestion and absorption of nutrients thereby optimizing fullness,reducing food intake and limiting insulin response in pre- and post-menopausal women.

DETAILED DESCRIPTION:
This study is designed to gain a better understanding of meal viscosity and the utility of dietary sources of viscous polysaccharide fibers to modulate postprandial metabolic and satiety mechanisms in pre- and post- menopausal overweight women in order to optimize acute metabolic responses to meals as well as most favorably affect appetite, food intake and overall body weight control.

Objectives of this study include:

1. To investigate the effects of viscous polysaccharide type fibers in a meal on postprandial intestinal-phase mechanisms of satiety [eg., cholecystokinin (CCK)] and meal-associated metabolic (eg., glucose, insulin, triglyceride) response patterns to low glycemic index (GI), fiber-controlled preload meals compared to a low fiber, high GI meal in overweight pre- and post- menopausal women.
2. To characterize the subjective and behavioral satiety responses to study-specific preload meals varying in viscous fiber content as well as determine the relationship of these satiety responses to the preload-associated physiological responses in overweight pre- and post- menopausal women.
3. To examine the influence of menopausal status of overweight women on the physiological, subjective and behavioral responses to study preloads.

The study is a randomized, 3-arm, 6-sequence, within-subjects, crossover, treatment-controlled study utilizing a repeated measures, multiple sampling paradigm to evaluate the metabolic and satiety response pattern to low glycemic index (GI) fiber-controlled preload treatments differing in viscous fiber content compared to a high GI preload meal.

The study will test 3 isocaloric treatment preloads in relatively healthy overweight, mildly obese, pre- and post- menopausal women. Preload meals will be prepared as breakfast meals using muffins and yogurt beverage / shake as the base for which glycemic index (GI) of the meal, including fiber / viscous fiber content, will be manipulated. All preloads have been matched as close as possible on sensory qualities as well as macronutrient composition, fiber and energy content and volume.

The 3 treatments will include as fiber source either viscous polysaccharide fiber source, eg., psyllium husk, and insoluble non-viscous producing fiber source, eg., cellulose, respectively. These fibers are commercially available.

Preload meals will be prepared to contain about 1 kcal/g offered as a 600 kcal meal portion. The macronutrient distribution for fat, carbohydrate and protein will be 30%, 55% and 15% of energy, respectively. Fiber will be included at 2 levels: 2 g/100 kcal for the 2 fiber containing preload meals and no fiber for the high GI low fiber control. These levels of fiber are consistent with our previously studied breakfast meals and for the higher fiber meals, just above the recommended intake for adult Americans. Preload meals will be matched as closely as possible on micronutrients and sensory (palatability, sweetness, texture) quality.

Preload meals be provided under fasting conditions and consumed within 20 minutes. Subsequent food intake will be measured in lab at a test meal and then by food records at home thereafter.

Subjects will receive each preload meal in random order ~ 1 month apart in order to standardize cyclic phase within the pre-menopausal group. Each preload test session will include collection of food records and menstrual logs, in-lab preload and test meal consumption, multiple blood sampling and visual analog scale completion.

Blood sample collection and visual analog scale (VAS) completion will occur before (fasting, time 0) preload meal consumption and then at 20, 40, 60, 90, 120, 150, and 180 min thereafter. A test meal lunch will be offered 2.5 h post-preload meal consumption. Test meal will be provided ad libitum. Final two blood draws and satiety evaluation will occur after lunch (210 and 240 minutes).

Blood will be measured for glucose, insulin, triglycerides and CCK at the specific time periods listed above. Occuring at the same time period, the subject will complete the VAS, a validated method for assessing subjective measures of appetite. Subjects will also rate the preload meals using the VAS on a number of sensory qualities to assess palatability.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years or older
* Unrestrained [score ≤ 10] on the Eating Inventory (EI) questionnaire
* Pre-menopausal with spontaneous cycle
* Post-menopausal ≥ 12 month without menstruation
* Body mass index (BMI) of either 25 to 33 kg/m2, inclusive

Exclusion Criteria:

* Pregnant and lactating
* Smoking
* Allergies or intolerances to foods consumed in the study
* Fasting glucose > 110 mg/dL
* Active modification to diet or exercise patterns to gain or lose weight in previous 60 days
* Unstable body weight (fluctuations of ≥ 5 kg in 60 day period)
* Excessive exercisers or trained athletes
* Taking any medications that would affect appetite or have a current or past (previous 1 year) medical condition that may interfere with any of the outcomes of this study.
* Hormonal therapy (ie., estrogen, progesterone)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-08-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
To investigate the effects of viscous polysaccharide fibers on postprandial satiety. | 0, 20, 40, 60, 90, 120, 150, 180, 210, 240 minutes
  Effect of Different Treatments on Cholecystokinin (CCK) Concentration
To investigate the effects of viscous polysaccharide fibers on postprandial meal-associated metabolic response patterns. | 0, 20, 40, 60, 90, 120, 150, 180, 210, 240 minutes
  Plasma glucose, insulin, and triglyceride concentrations measured by Randox Clinical analyzer

SECONDARY OUTCOMES:
To characterize the subjective and behavioral satiety responses to study-specific preload meals varying in viscous fiber content as well as determine the relationship of these satiety responses to the preload-associated physiological responses. | 0, 20, 40, 60, 90, 120, 150, 180, 210, 240 minutes
  Satiety measured by Three-Factor Eating Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, MS, PhD, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almiron-Roig E, Chen Y, Drewnowski A. Liquid calories and the failure of satiety: how good is the evidence? Obes Rev. 2003 Nov;4(4):201-12. doi: 10.1046/j.1467-789x.2003.00112.x. PMID 14649371
- [Background] Anderson GH, Moore SE. Dietary proteins in the regulation of food intake and body weight in humans. J Nutr. 2004 Apr;134(4):974S-9S. doi: 10.1093/jn/134.4.974S. PMID 15051857
- [Background] Burton-Freeman B. Sex and cognitive dietary restraint influence cholecystokinin release and satiety in response to preloads varying in fatty acid composition and content. J Nutr. 2005 Jun;135(6):1407-14. doi: 10.1093/jn/135.6.1407. PMID 15930445
- [Background] Schneeman BO, Burton-Freeman B, Davis P. Incorporating dairy foods into low and high fat diets increases the postprandial cholecystokinin response in men and women. J Nutr. 2003 Dec;133(12):4124-8. doi: 10.1093/jn/133.12.4124. PMID 14652359
- [Background] Burton-Freeman B, Davis PA, Schneeman BO. Plasma cholecystokinin is associated with subjective measures of satiety in women. Am J Clin Nutr. 2002 Sep;76(3):659-67. doi: 10.1093/ajcn/76.3.659. PMID 12198015
- [Background] Burton-Freeman B, Davis PA, Schneeman BO. Interaction of fat availability and sex on postprandial satiety and cholecystokinin after mixed-food meals. Am J Clin Nutr. 2004 Nov;80(5):1207-14. doi: 10.1093/ajcn/80.5.1207. PMID 15531667